CLINICAL TRIAL: NCT04000646
Title: Impact of a Breath-controlled Video Game App on Preoperative Anxiety, Induction Behavior and Parent Experience: A Randomized Controlled Trial
Brief Title: Impact of a Breath-controlled Video Game App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-0654
Record Dates: First submitted 2019-06-23; First posted 2019-06-27 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anxiety Acute
Keywords: anxiety, children
MeSH Terms: conditions — Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Other): Standard care non-pharmacologic interventions during anesthesia induction
  Interventions: Other: standard care
- breath-controlled app (Experimental): breath-controlled app and custom-designed tablet (equipped with a breathing sensor)
  Interventions: Other: breath-controlled app

INTERVENTIONS:
Other: standard care — standard care non-pharmacologic interventions during anesthesia induction
  Arms: standard care
Other: breath-controlled app — breath-controlled app and custom-designed tablet (equipped with a breathing sensor)
  Arms: breath-controlled app

SUMMARY:
The proposed research study will assess the impact of a newly developed, breath-controlled app and custom-designed tablet (equipped with a breathing sensor) on the patient and parent's preoperative anxiety and anesthesia induction experience.

DETAILED DESCRIPTION:
Aim 1: Determine whether induction distress differs between patients using the breathing-controlled app and those using standard care interventions: The investigators will measure patient compliance with induction using the Child Induction Behavioral Assessment (CIBA). The investigators predict that patients using the breathing-controlled app will demonstrate significantly better induction compliance. Older children (ages 6-8) are typically more cooperative with induction than younger children (ages 3-5 years). Both age groups will be studied to determine whether there are age-related differences impacting receptiveness to the app.

Aim 2: Compare patient anxiety between the breath-controlled app and control group. The investigators will measure child preoperative anxiety (modified Yale Preoperative Anxiety Scale, the "mYPAS-SF"). The investigators predict there will be significantly lower anxiety (mYPAS-SF) during induction for children in the breath-controlled app group.

Aim 3: Compare parent anxiety between the breath-controlled app and control group. The investigators will measure parental anxiety using the Visual Analog Scale for Anxiety, the "VAS-A". The investigators predict there will be significantly lower anxiety (mYPAS-SF) during induction for parents in the breath-controlled app group.

Aim 4: Determine overall family satisfaction with the induction experience. A survey will be administered to assess satisfaction levels with induction behavioral interventions and determine whether these scores differ between the intervention and standard care group. The investigators predict that satisfaction scores will be higher in the intervention group than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Same Day Surgery department at CCHMC Liberty campus
* Outpatient or 23 hour admission
* Any surgery or procedure under anesthesia
* Ages 3 to 8 years
* Male or female
* Any ethnicity
* American Society of Anesthesiologists (ASA) physical classification status I or II
* Patient has never had a prior anesthetic
* Family and participant communicate primarily in English & signed English anesthesia consent
* Normal neurocognitive development
* Patient is undergoing inhalation induction using an anesthesia mask
* Parent/guardian is present for induction
* Patient does not receive a premedication for anxiety

Exclusion Criteria:

* Neurocognitive delays
* Developmental delays/Behavioral diagnoses, such as (but not limited to) ADHD, Autism, Oppositional defiant disorder, Obsessive Compulsive Disorder, Anxiety disorder
* Patient takes medications routinely for behavioral issues
* Tracheostomy
* Inpatient or planned >23 hour admission

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Primary aim (induction distress) | During anesthesia induction
  Induction distress (Child induction behavioral assessment tool, the "CIBA"), scored by reviewing behavioral descriptions of 3 categories, "Smooth, "Moderate", or "Difficult"

SECONDARY OUTCOMES:
Secondary aim (anxiety) | Child preoperative anxiety (in Same Day Surgery) and anxiety during anesthesia induction (measured during induction)
  Child anxiety (modified Yale Preoperative Anxiety Scale, the "mYPAS-SF"), scored 23-100, 100 = highest anxiety score
Secondary aim (anxiety) | Parental preoperative anxiety (in Same Day Surgery) and anxiety during anesthesia induction (measured immediately after induction)
  Parental anxiety (Visual Analog Scale for anxiety, the "VAS-A"), scored 0-100, 100 = highest anxiety score
Secondary aim (satisfaction) | Immediatly after anesthesia induction
  Family satisfaction with the induction experience (survey, Likert scale, 1= poor; 10 = excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Abby Hess, DNP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No